CLINICAL TRIAL: NCT03175497
Title: A Phase I Study to Evaluate Safety, Tolerability and Pharmacokinetics of Telatinib, a Selective Inhibitor of the Vascular Endothelial Growth Factor (VEGF) Receptor, in Adult Chinese Patients With Advanced Solid Tumors
Brief Title: Telatinib Safety and Pharmacokinetics Study in China Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taizhou EOC Pharma Co., Ltd. (Industry)
Collaborators: Fountain Medical Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOC315001
Record Dates: First submitted 2017-05-25; First posted 2017-06-05 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor, Adult
Keywords: Gastric Cancer, VEGFR inhibitor
MeSH Terms: conditions — Stomach Neoplasms | interventions — telatinib

STUDY DESIGN:
Intervention Model Description: This study is comprised of two stages. The 1st stage will follow the traditional 3+3 dose-escalation design in patients with advanced solid tumor The 2nd phase will be conduced in Gastric cancer patients, primarily for PK data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telatinib mesylate treatment arm (Experimental): Open label, single arm trial. For the 1st phase: three cohorts, and each with 3-6 solid tumor patients who will be treated with telatinib at predetermined dose: 600 mg bid, 900 mg bid, or 1200 mg bid, respectively.
  For the 2nd phase, one cohort with 12 GC patients who will be treated with telatinib at 900 mg bid
  Interventions: Drug: Telatinib Mesylate

INTERVENTIONS:
Drug: Telatinib Mesylate — Telatinib mesylate tablets will be administrated twice a day orally
  Other Names: BAY 57-9352, TEL0805, EOC315

SUMMARY:
The purpose of this China Phase I bridging study is to to evaluate the safety, tolerability and pharmacokinetic profile of telatinib in China patients with advanced solid tumor

DETAILED DESCRIPTION:
This is an open-label, nonrandomized, phase I, escalating dose study to evaluate the safety, tolerability and pharmacokinetic profile of telatinib. .

This study is comprised of two stages. The 1st stage follows the traditional 3+3 dose-escalation design. Telatinib mesylate tablets will be administrated orally to patient twice daily at a starting dose of 600 mg bid. Patients will be successively enrolled into three cohorts from low-dose to high-dose (600 mg bid, 900 mg bid, and 1200 mg bid). For each cohort, patient will be first enrolled for single-dose PK and safety observation. After one-day interval, patient will then be resumed for a 21-day continuous treatment to assess safety, tolerability and PK profile with multiple dosing.

The dose-limiting toxicity (DLT) observation period will be 23 days, starting from the first day of single dosing till the end of the 21-day continuous treatment.

If first 3 subjects at a dose level complete a cohort without experiencing any DLT, subjects for the next higher cohort will be recruited. If 1 of the first 3 subjects experiences DLT, then up to three additional subjects (total up to six subjects) will enrolled at that dose level. If more than 2 patients at a dose level experienced DLT, dose escalation will be halted. And the dose level will be declared the toxic dose. The MTD is defined as the previous (lower dose) dose level.

If MTD is not observed even at 1200 mg bid, dose-escalation will not be continued.

ELIGIBILITY:
Inclusion Criteria

For inclusion in the study patients should fulfil the following criteria:

1. Provision of informed consent prior to any study specific procedures.
2. ≥ 18 and ≤ 70 years of age
3. For the 1st phase: histological or cytological confirmed solid malignant tumors in advanced stage, standard regimen failed or intolerable, or no standard regimen available For the 2nd phase: histological or cytological confirmed gastric cancer in advanced stage.
4. ECOG performance status of 0-1
5. Life expectancy of more than 12 weeks
6. Patients must have adequate organ and bone marrow function as defined by the following laboratory results.

   1. Neutrophil > 1.5 × 10^9/L
   2. Platelets >100 × 10^9/L
   3. Alkaline phosphatase ≤2 times the upper limit of normal (ULN)
   4. Prothrombin time (PT), international normalized ratio (INR), and partial thromboplastin time (APPT) < 1.5 times ULN
   5. Hemoglobin ≥ 9 g/dL.
   6. Creatinine ≤ 1.5 times the upper limit of normal (ULN) for the institution or Creatinine clearance ≥ 60 ml/min
   7. Total bilirubin ≤ 1.5 times ULN
   8. Aspartate transaminases (AST/SGOT) or alanine transaminase (ALT/SGPT) ≤ 2.5 times ULN. In HCC patients, those two values should be < 5 times ULN
   9. Urine protein <2+; if urine protein ≥ 2+, 24-hour urine protein quantity must ≤ 1g
7. Patients must be able to swallow tablets, not spit out the drug, and without malabsorption
8. Patients must NOT suffer from medical or psychiatric conditions that would interfere with protocol compliance, the ability to provide informed consent, or assessment of response or anticipated toxicities.

Exclusion Criteria:

Patients should NOT enter the study if any of the following exclusion criteria are fulfilled:

1. Patients have known central nervous system metastasis except patients who have terminated steroid treatment for brain metastasis or spinal cord compression with remain disease stable for at least 1 month. (a MRI is not required to rule out brain metastases unless there is clinical suspicion)
2. Patients with diagnosed lymphoma
3. Patients receiving the following therapy or treatment prior to enrollment:

   1. Mitomycin C or nitroso urea within ≤ 6 weeks immediately prior to C1D1; anticancer drugs, chemotherapy, radiation or immunotherapy within ≤ 4 weeks immediately prior to C1D1, or have not recovered from the prior anticancer therapy that was received 4 weeks ago (Anticancer drug therapy is defined as any drug or drug combination that have demonstrated anticancer activities, and the purpose of application is to directly or indirectly influence cancer. Patients who have ever received the following therapies can be enrolled: adjuvant chemotherapy, chemotherapy, immunotherapy or steroid therapy for metastatic diseases)
   2. Autologous bone marrow transplantation or stem cell therapy within ≤ 4 weeks immediately prior to C1D1
   3. Biological regulators, such as granulocyte colony stimulating factors (G-CSF)
4. Patients who need to take anticoagulant medications throughout the study (such as heparin, warfarin, clopidogrel and aspirin)
5. Patients who have a history of heart disease: NYHA III or IV grade of congestive heart failure, coronary artery disease; or have been hospitalized due to heart failure, atrial fibrillation, or atrial flutter within ≤ 3 months immediately prior to C1D1
6. Patients who suffer from ≥ grade 2 myocardial ischemia and myocardial infarction; poorly controlled cardiac arrhythmia, including QTc : men ≥ 450 ms, women ≥ 470 ms (patients are only allowed to receive beta blockers or dioxin)
7. Patients who suffer from hypertension (systolic blood pressure > 140 mmHg or diastolic pressure is 90 mmHg) that cannot be controlled by receiving ≤ two types of antihypertensive drugs
8. Patients who have a medical history of HIV infection, active hepatitis B or hepatitis C infection.
9. Patients who suffer from severe unhealed damage, bleeding, ulcer and fracture
10. Patients who have evidence of severe or poorly controlled systemic disease (e.g., severe liver damage, severe kidney damage, poorly controlled diabetes and acute infection), or unstable current diseases, or decompensated respiratory or cardiac disease (baseline LVEF < 55%), or peripheral vascular disease (including diabetic vascular disease);
11. Patients who have gone major surgery ≤ 4 weeks immediately prior to C1D1, including but not limited to hip or knee replacement, or spinal cord injury
12. Patients who have a medical history of venous thromboembolism
13. Patients who suffer from seizure that needs to be controlled by drug
14. Patients who have the high risk of developing coagulation, and are defined as those who meet any two of the following criteria

    1. Platelets >300 × 10^9/L
    2. PT reduction >3s (8.8-13.8s)；
    3. APPT reduction >3s (24.9-36.8s)
    4. Fibrinogen (FIB) > 0.5 g/L
    5. D-dimer > 300 μg/L
15. Patients who have a medical history of organ transplantation
16. Patients who have ever received telatinib treatment
17. Patients who have received any investigational agent within ≤ 4 weeks immediately prior to C1D1 or plan to receive other investigational agent during the course of this study
18. Patients who have known or suspected allergies to telatinib mesylate tablet, its recipients, and drugs of the similar class
19. Women who are breast-feeding, or have positive results of serum pregnancy test within ≤ 7 days immediately prior to C1D1, or sexually active males and pre/perimenopausal women who do not agree to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study and for 3 months after discontinuation of therapy
20. Patients who suffer from medical or psychiatric conditions that would interfere with protocol compliance, the ability to provide informed consent, or assessment of response or anticipated toxicities.
21. Patients are not suitable for the enrollment based on the judgment of Investigators
22. People who are involved in the planning and conduct of the study (applies to both Eddingpharm. LTD staff and staff at the investigational site).

    Patients with advanced GI tumor in the 1st phase and all patients in the 2nd phase should be excluded from enrollment if any of the following criteria is met:
23. Patients who ever suffer from active gastrointestinal bleeding or occult blood (++) within ≤ 4 weeks immediately prior to C1D1
24. Patients who suffer from occult blood (+) and the enteroscopy results assessed by Investigator with the potential of causing gastrointestinal bleeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity, incidence of treatment-emergent adverse events | single dose, and twice daily continuous dosing for 21 days
  Other safety and tolerability parameters including 12-lead ECG, vital signs, blood pressure/pulse, temperature, physical examination, laboratory parameters (hematology, blood biochemistry, coagulant examination, thyroid function test and urine test), and ECOG score.

SECONDARY OUTCOMES:
Cmax | single dose, and twice daily continuous dosing for 21 days
  Peak Plasma Concentration
AUC | single dose, and twice daily continuous dosing for 21 days
  Area under the plasma concentration versus time curve

OTHER OUTCOMES:
Explore potential predictive and prognostic biomarkers associated with telatinib treatment | prior to treatment and after 21-day treatment
  Plasma level of soluble VEGFR2

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University, Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No